CLINICAL TRIAL: NCT04341740
Title: Investigating Marrow Infiltrating Lymphocytes as a Source of Adoptive Cellular Therapy in Renal Cell Carcinoma and Urothelial Carcinoma
Brief Title: Investigating Marrow Infiltrating Lymphocytes in Renal Cell Carcinoma
Acronym: WindMIL-001
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study funding was withdrawn.
Sponsor: University of Oklahoma (Other)
Collaborators: WindMIL Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OI-SCC-WINDMIL-001
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Renal Cell Carcinoma; Urothelial Carcinoma
Keywords: marrow infiltrating lymphocytes
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Transitional Cell

STUDY DESIGN:
Intervention Model Description: Patients enrolled on this study in either the Renal Cell Carcinoma cohort or the Urothelial Carcinoma cohort will undergo the same procedures of bone marrow aspiration and blood draw.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Renal Cell Carcinoma or Urothelial Carcinoma Patients (Experimental): Patients in both cohorts (RCC or UC) will undergo bone marrow aspiration under conscious sedation to withdraw 60 mL bone marrow aspirate and 75 ml of peripheral blood sample.
  Interventions: Procedure: Bone Marrow Aspirate

INTERVENTIONS:
Procedure: Bone Marrow Aspirate — bone marrow aspiration

SUMMARY:
The purpose of this research is to collect health-related information as well as bone marrow and blood specimens to determine if a new form of treatment for patients with kidney and bladder cancer may be possible.

DETAILED DESCRIPTION:
This research will collect specimens from the bone marrow and blood to determine if a new treatment for kidney or bladder cancer may be possible. This research study will collect a bone marrow sample as well as a blood sample.

Participation in the research study will last approximately 60 days which includes time to determine if the patient is eligible to participate in the study, perform the research procedures and follow-up with the patient following the research procedures to determine if they are experiencing any side effects. Participation will end approximately 30 days following the bone marrow collection.

The bone marrow and blood samples will be collected from all patients in both cohorts only at a single time point, after they have been enrolled on the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically-confirmed, locally advanced unresectable or metastatic RCC (cohort A) or UC (cohort B).
* ECOG performance status of ≤1
* Adequate bone marrow function:

  * Platelet count ≥ 100 × 10^9/L
  * ANC ≥ 1.0 ×10^9/L
  * Lymphocyte count ≥ 0.5 ×10^9/L
* Willingness to undergo bone marrow aspiration (BMA)

Exclusion Criteria:

* Prior hematopoietic stem cell transplantation
* Prior radiation to the pelvic region
* Use of systemic corticosteroids within 28 days of BMA
* History of another primary malignancy that has been diagnosed or required therapy within the past 2 years (except completely resected basal cell and squamous cell skin cancer, curatively treated localized prostate cancer, and completely resected carcinoma in situ of any site).
* Presence of an autoimmune disease (e.g., rheumatoid arthritis, multiple sclerosis, systemic lupus erythematosis) requiring active systemic treatment. If the autoimmune disease has been treated, it must be stable clinically. (Hypothyroidism without evidence of Grave's disease or Hashimoto's thyroiditis is not considered an exclusion criterion.)
* Pregnant females as documented by a serum beta human chorionic gonadotropin (β-hCG) pregnancy test consistent with pregnancy, obtained within 21 days of BMA
* Infection requiring treatment with antibiotics, antifungal, or antiviral agents within 7 days of BMA
* Known diagnosis of HIV or CMV infection or active viral hepatitis
* Administration of hematopoietic growth factor support within 14 days before bone marrow aspiration
* Chemotherapy administration within 28 days of BMA
* Unwilling or unable to comply with the protocol
* Prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the Investigator's opinion, could affect the safety of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with successful isolation and ex-vivo expansion of MILs | 30 days
  A successful expansion will be greater than or equal to 50% viable and greater than or equal to 50% CD3 positive.

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Tripathi, MD, Principal Investigator — University of Oklahoma
Locations (1):
- Stephenson Cancer Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No